CLINICAL TRIAL: NCT05955807
Title: Tracking Suicidal Ideation and Factors That Influence it in High-risk Patients After Discharge From Psychiatric Acute Wards. An Ambulatory Momentary Experience-sampling Study
Brief Title: Momentary Assessment.Tracking Suicidal Ideation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: Vestreviken
Record Dates: First submitted 2023-04-21; First posted 2023-07-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-08

CONDITIONS: Suicide Risk; Suicide Ideation; Suicide Prevention; Ecological Momentary Assessment; Suicide Attempt
MeSH Terms: conditions — Suicide Prevention; Suicide, Attempted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized due to severe risk of suicide: This is an observational study that focus on patients wellbeing and life-experience in the discharge period after a stay in psychiatric care due to severe risk of suicide. Patients will be treated according to usual pratice in clinical care

SUMMARY:
The goal of this observational study is to increase the knowledge base about fluctuations in suicide ideation and its association with relational and contextual factors after hospital discharge in patients with high risk of suicide. Patients hospitalized due to severe risk of suicide (recent suicide attempt or due to acute suicidality) are invited to participate in the study. Researchers will investigate how psychological, relational and contextual factors trigger as well as protect against escalating suicide ideation in this period in the post discharge period. Information will be retrieved from multiple sources (eg. by Ecological Momentary Assessment Method (EMA), regular patient interviews and questionnaires in addition to information from Electronic Patient Registry) to; a) delineate fluctuations in suicide ideation, b) identify factors that are associated with/ influence suicide ideation in the EMA assessment period, c) explore associations with relational and contextual measures during EMA assessment, d) generate profiles for subgroups and investigate how participants experience and evaluate their participation and completion of the EMA assessment protocol.

DETAILED DESCRIPTION:
Suicide risk is high amongst patients in mental health services in the postdischarge period (Large & Kapur, 2018; Chung et al 2019). However, our current knowledge and understanding does not help us in preventing suicide as an outcome. It is not possible to predict suicide in high risk populations, and- more importantly- we also are not able in any efficient way to discriminate between those who are at higher risk for suicide and those who are in less high risk of suicide in this population (Franklin et al 2017, Large, 2018).

The most limiting feature of current procedures for suicide risk assessment is their very broad based, coarse characteristics, with a notable lack of incorporated knowledge of how ongoing daily life experiences influence suicide risk. If clinical judgments on suicide risk are to reach a higher level of certainty, this can only be achieved by addressing the specific, proximal factors that maximally relevant to the patients and their situation (Nock et al, 2009).

The field of suicidology needs to determine how, when and for whom continued life suffering after discharge are accompanied by increased suicidal risk. Further important tasks are to identify the post-discharge factors that protect these patients. In this context, the aim is to increase the knowledge base about fluctuations in suicide ideation and its association with relational and contextual factors after hospital discharge in suicide attempters and patients hospitalized to psychiatric institutions due to severe suicide risk. Moreover, the researchers aim to determine "profiles" of such associations for different patient subgroups. These profiles of associations will be regressed against the presence vs absence of novel suicide risk behavior including possible self-harm and suicide episodes as a subsequent follow up point months later. Hence, the core data from the project will be seen in relation to both suicidal thoughts and subsequent suicidal behavior.

Below, four Research Questions (RQ) including specific hypotheses are described.

RQ1: Delineate fluctuations in suicide ideation

1. In the overall patient group considered together, suicide ideation (degree and endurance) will fluctuate markedly within a day and over the assessment period
2. Patient characteristics and patient subgroups can be identified, with different fluctuations in suicide ideation, including absence of suicide ideation at most time points, stable levels of suicide ideation, highly fluctuating levels, and duration of suicide ideation

RQ2: Identify factors that are associated with/ influence suicide ideation in the EMA assessment period

1. Associations with patient characteristics at baseline: Overall, suicide ideation will be at higher levels and fluctuate more profoundly, in individuals with high baseline scores on the following: i) psychological pain, stress, agitation or inner turmoil, hopelessness and self-hate, ii) high severity of their recent suicide attempt, and iii) high levels of depression and general symptom severity, in addition to (iv) in individuals who live socially isolated/ alone versus those who live together with a partner or family
2. Associations with relational and contextual measures during EMA assessment:

i. Suicide ideation will be relatively high as well as enduring in times of i) psychological pain, stress, agitation or inner turmoil, hopelessness and self-hate, ii) interpersonal conflict, iii) when they are alone or with friends and negative feelings dominate over positive feelings, and iv) when perceived control over thoughts is low ii. Suicide ideation will be absent when i) patients are in relations with other people and (ii) when they experience positive feelings

RQ3: Generate profiles for subgroups

1. Based on findings for RQ1-RQ3, different profiles of associations between suicide ideation and other EMA measures can be delineated for different subgroups of patients, and that can be reliably linked to patient characteristics at baseline
2. Explore differences in suicide ideation and related cognitions/ other EMA measures in the group with and without a suicide attempt
3. High risk profiles can be identified by linking associations between suicide ideation and other EMA measures to subsequent suicide ideation, symptom severity, self-harm, and/ or suicide attempts at 3 weeks and 3 months follow-up

RQ4: How do participants experience and evaluate their participation and completion of the EMA assessment protocol?

This is a longitudinal observational study. The researchers will adopt the method of Ecological Momentary Assessment to assess how participants cope in the postdischarge period. Participants will receive 5 surveys daily in the first 10 days after leaving the hospital. Additionally, participants will meet to three research interviews; baseline interview before discharge from the hospital, after three weeks and after three months

Measures (see section for outcome measures)

The multi-level EMA data (assessments nested within days and participants) will be analyzed in mixed effect regression models, focusing on linear changes in suicidal ideation over time and on how this is associated with independent variables. To estimate within-subject and between-subject variation, the patient identifier and time will be the random variables in the mixed effect model. In the random part of the mixed model, the residual is the estimate for within-subject variation. In prospective analyses (from T to T+1), time-lagged variables will be used as predictors. Data will be centered prior to analysis, with centering model based on the hypothesis to be tested.

Statistical power in multilevel data depends on number of both individuals and assessments.

With 5 daily assessments over 10 days in 50 participants, power is 100% to detect large effect sizes and 80% to detect medium effect sizes (as modeled by Power Curves for Multi-level Studies (shinyapps.io).

References- Chung, D., et al., Meta-analysis of suicide rates in the first week and the first month after psychiatric hospitalisation. BMJ Open, 2019. 9(3): p. e023883.

Franklin, J.C., et al., Risk factors for suicidal thoughts and behaviors: A meta-analysis of 50 years of research. Psychol Bull, 2017. 143(2): p. 187-232.

Large, M. and N. Kapur, Psychiatric hospitalisation and the risk of suicide. Br J Psychiatry, 2018. 212(5): p. 269-273.

Large, M., The role of prediction in suicide prevention. Dialogues Clin Neurosci, 2018. 20(3): p. 197-205.

Nock, M.K., M.J. Prinstein, and S.K. Sterba, Revealing the form and function of self-injurious thoughts and behaviors: A real-time ecological assessment study among adolescents and young adults. J Abnorm Psychol, 2009. 118(4): p. 816-27.

ELIGIBILITY:
Inclusion Criteria

1. Patients hospitalized with a recent suicide attempt or
2. Patient hospitalized due to severe risk of suicide

Exclusion Criteria

1. Active psychosis
2. Developmental disorders
3. Intellectual disability
4. Poor norwegian acquisition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in psychiatric care in Norway are characterized by high symptom severity and comorbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Fluctuations in suicide ideation | 10 day Ecological Momentary Assessment-registrations
  Fluctuations in Suicide Ideation and related variables (eg. "I wish to live", "I wish to die" "I think about taking my own life", "I feel hopeless". Questions are rated on a Likert scale (1-5). Participant will answer questions on their mobile-phone 5 times each day for 10 days.

SECONDARY OUTCOMES:
Suicidal behaviors | Baseline, 3 weeks after discharge, and then again 3 months after discharge
  The Suicide Attempt Self-injury Count (SASIC-interview)
General symptom severity | Baseline and 3 months
  Outcome Questionnaire 45 (Likert scale 0-4, 45 questions, where high scores refers to high symptom severity)
Depression | baseline
  Patient Health Questionnaire-9 (Likert scare 0-3. 9 questions, where high scores indicate higher symptom severity)
Experience with using the EMA app | 3 weeks
  User Satisfaction Survey on patient experience with EMA-assessment (1-5, 6 questions where higher scores indicate that the participant agrees more to the statement)
Suicide Ideation | Baseline, 3 weeks, 3 months
  Beck Scale for Suicide Ideation- Current (0-2, 19 questions. Higher scores indicate more severe suicide ideation)
Suicide ideation | Baseline, 3 weeks, 3 months
  Suicide Status Form-IV (1-5, where higher scores indicate more symptoms)
EMA questionnaire protocol | 10 day intensive tracking og experiences
  26- 28 questions covering; mood, suicide ideation, significant recent events, context and actions. Likers scale questions are scaled from 1-5 or 1-7, where higher scores indicate higher intensity.

OTHER OUTCOMES:
Baseline characteristics/ descriptive variable/ diagnostic group | baseline
  The Mini Psychiatric Interview (MINI)
Psychological diagnostic group | 3 weeks
  Structured Clinical Interview 5- Personality Disorder (SCID-5-PF)
general patient demographics | baseline and 3 months
  (previous and current treatment history, number of rehospitalizations during the project period, work status, social setting aso

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Research and Delvelopment, Mental health and Addiction, Vestre Viken Hospital Trust, Drammen, Norway

IPD SHARING:
Plan to Share IPD: Undecided